CLINICAL TRIAL: NCT00985595
Title: Quality Community Services for Adolescent Drug Abuse
Brief Title: Learning Effective Approaches to Prevention
Acronym: CASALEAP
Status: Completed | Type: Observational
Sponsor: The National Center on Addiction and Substance Abuse at Columbia University (Other)
Responsible Party: Principal Investigator, Aaron Hogue, Director of Adolescent and Family Research, The National Center on Addiction and Substance Abuse at Columbia University
Other Study IDs: 165; 1R01DA019607-01 (NIH)
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Adolescent Substance Abuse
Keywords: Adolescent; substance abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of the study is to test the effectiveness, implementation quality, and cost effectiveness of family-based treatment services for adolescent substance abuse delivered in an agency setting.

DETAILED DESCRIPTION:
Despite the success of family-based ecological interventions (FBEI) in controlled trials, this highly promising services approach has not been tested under pure field conditions with ASA populations. Controlled effectiveness research invariably enhances training, supervision, and service delivery conditions in partnering sites in an effort to ensure treatment adherence and consistency. An alternative strategy for advancing dissemination science is rigorous naturalistic research on community clinics that already implement evidence-based practices in the course of routine care. The proposed study will follow this "bottom up" strategy by investigating the quality and impact of ASA services delivered by front-line therapists in a community-based mental health center that already features FBEI as the routine standard of care. The study will use a randomized design to compare naturalistic FBEI services to services as usual (SAU) for ASA. Participants (N = 260) will be recruited from local high schools, enrichment programs, and juvenile justice programs. Eligible adolescents will meet ASAM criteria for outpatient treatment. The SAU condition will contain the three most common service venues for ASA in urban communities: hospital-based ambulatory mental health clinics, drug counseling/addictions specialty clinics, and community mental health centers. The primary aims of the study are to examine the effectiveness of FBEI versus SAU and to compare the strength of FBEI adherence and outcomes to performance benchmarks set during a previous FBEI Stage II efficacy trial. The secondary aims are to compare cost effectiveness, services utilization, and consumer satisfaction in FBEI versus SAU. A multitrait, multimethod assessment design will include adolescent and parent interviews at baseline and 3, 6, and 12 months follow-up. Cost and service utilization data will be collected from self report and from provider agencies in both conditions. The study will yield the first evidence on whether a widely endorsed treatment approach for ASA is potent and feasible in real-world conditions and superior to SAU in outcomes and cost-benefit. An important secondary yield will be increasing the scarce knowledge base on commonly practiced community approaches in the SAU condition.

ELIGIBILITY:
Inclusion Criteria:

1. ages 13 and 17,
2. have a caregiver willing to participate in treatment,
3. meet ASAM criteria for outpatient or intensive outpatient substance abuse treatment,
4. not receiving any other behavioral treatment, and
5. have public or private health benefits that meet standard community clinic registration requirements.

Exclusion Criteria:

1. mental retardation,
2. pervasive developmental disorder,
3. medical or psychiatric illness requiring hospitalization,
4. current psychotic features, or
5. current suicidality (Ideation + Plan + High Intention).

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adolescents screened for symptoms of substance abuse/dependence, and their families, will participate in the study. Participants will include 260 male and female adolescents who complete the enrollment process, meet eligibility criteria, and consent to be randomized into one of two study conditions. Youth will be referred primarily from two sources: juvenile justice agencies and local schools/community programs. Based on the demographics of adolescents currently participating in partner sites, youth are likely to be predominantly male (69%), Hispanic (68%), and African American (32%). Families are generally low income from disadvantaged neighborhoods, with high rates of family mental health and substance use problems.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2006-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The primary aims of the study are to examine the effectiveness of FBEI versus SAU and to compare the strength of FBEI adherence and outcomes to performance benchmarks set during a previous FBEI efficacy trial. | 3, 6, 12 months after baseline

SECONDARY OUTCOMES:
The secondary aims are to compare cost effectiveness, services utilization, and consumer satisfaction in FBEI versus SAU. | 3, 6, 12 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Hogue, Ph.D., Principal Investigator — The National Center on Addiction and Substance Abuse at Columbia University
Locations (1):
- The National Center on Addiction and Substance Abuse at Columbia University, New York, New York, United States

REFERENCES:
- [Derived] Mattos LA, Schmidt AT, Henderson CE, Hogue A. Therapeutic alliance and treatment outcome in the outpatient treatment of urban adolescents: The role of callous-unemotional traits. Psychotherapy (Chic). 2017 Jun;54(2):136-147. doi: 10.1037/pst0000093. Epub 2016 Nov 10. PMID 27831697